CLINICAL TRIAL: NCT02133547
Title: Determination of Normal Values of Nasal Nitric Oxide Measured With the NIOX MINO Analyzer in Adults: a Pilot Study
Brief Title: Determination of Normal Values of Nasal Nitric Oxide in Adults
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr. Romain Lazor, MD, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CHUV-PNE-nNO-01
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Normal Values of Nasal Nitric Oxide in Healthy Adults
Keywords: Nitric Oxide; Nose; Healthy Volunteers; Kartagener Syndrome; Primary Ciliary Dyskinesia
MeSH Terms: conditions — Kartagener Syndrome; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary ciliary dyskinesia (PCD) is a rare genetic disorder characterized by impaired airway mucociliary clearance leading to recurrent respiratory infections, bronchiectasis and eventually respiratory insufficiency. Diagnosis of PCD is difficult and relies on complex methods which are not widely available (1).

Nasal nitric oxide (nNO) is reduced in PCD patients as compared to normal subjects, and nNO measurement has been proposed as a non-invasive screening tool for PCD. However, nNO measurement techniques are not standardized and reference values are lacking (2, 3).

The NIOX MINO is a handheld analyzer developed for the non-invasive measurement of exhaled NO (eNO) in asthmatics. Measurement of nNO with the NIOX MINO has been reported in only few studies (4-6), which mainly compared the NIOX MINO with others NO analyzers. However, no study attempted to establish reference values with the NIOX MINO in a large number of normal subjects.

One critical issue in nNO measurement is to avoid contamination of nasal air by exhaled alveolar air during nNO sampling. This can be obtained by either breath holding, or by a breathing technique allowing soft palate closure during sampling, such as mouth breathing again resistance. However, as sampling times with the NIOX MINO are long (2 minutes at a flow of 2 ml/min, and 45 seconds at a flow of 5 ml/min), these techniques may be difficult to apply.

In this pilot study, we will determine normal nNO values in 100 healthy men and women aged 20 to 70 years using 3 different breathing techniques:

1. breath holding during 45 seconds
2. mouth breathing through a fixed resistance (a straw), to create a small positive pressure in the oropharynx during expiration only
3. mouth breathing through a continuous positive airway pressure (CPAP) apparatus, which produces continuous soft palate closure during quiet spontaneous breathing, thus allowing long sampling times for nNO measurement.

This study will allow: 1) to determine whether nNO can be reliably measured with the NIOX MINO in adult normal subjects, 2) to identify the most reproducible breathing technique, 3) to determine normal values of nNO as measured by the NIOX MINO, and 4) to explore possible differences between genders and age groups.

References:

1. J.S.A. Lucas, W.T. Walker, C.E. Kuehni and R. Lazor. Primary ciliary dyskinesia. Eur Respir Mon. 2011; 54: 201-217.
2. ATS/ERS Recommendations for Standardized Procedures for the Online and Offline Measurement of Exhaled Lower Respiratory Nitric Oxide and Nasal Nitric Oxide, 2005. Am J Respir Crit Care Med 2005; 171: 912-30.
3. Marthin JK, Nielsen KG. Choice of nasal nitric oxide technique as first-line test for primary ciliary dyskinesia. Eur Respir J 2011; 37: 559-65.
4. Marthin JK, Nielsen KG. Hand-Held Tidal Breathing Nasal Nitric Oxide Measurement - A Promising Targeted Case-Finding Tool for the Diagnosis of Primary Ciliary Dyskinesia. PLoS ONE 2013; 8: e57262.
5. Weschta M, Deutschle T, Riechelmann H. Nasal fractional exhaled nitric oxide analysis with a novel hand-held device. Rhinology 2008; 46: 23-7.
6. Maniscalco M, Laurentiis G de, Weitzberg E, Lundberg JO, Sofia M. Validation study of nasal nitric oxide measurements using a hand-held electrochemical analyser. Eur J Clin Invest 2008; 38: 197-200.

ELIGIBILITY:
Inclusion Criteria:

* consent signed
* adult healthy subjects

Exclusion Criteria:

* current smoker
* history of asthma
* history of acute or chronic sinusitis
* history of nasal polyps
* upper airway infection in the past 3 weeks
* use of nasal corticosteroids in the past 3 weeks
* cleft palate
* history of uvulopharyngopalatoplasty
* history of neuromuscular disorder
* history of chronic respiratory disease, including cystic fibrosis and primary ciliary dyskinesia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
nitric oxide concentration in the air flowing through the nasal cavities | sampling time: 45 seconds
  The NIOX MINO is a handheld analyzer allowing determination of nitric oxide in an air sample. The sample is obtained non-invasively by breathing in the device through the mouth or nose.

CONTACTS AND LOCATIONS:
Overall Officials: Romain Lazor, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Respiratory Department Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Maniscalco M, de Laurentiis G, Weitzberg E, Lundberg JO, Sofia M. Validation study of nasal nitric oxide measurements using a hand-held electrochemical analyser. Eur J Clin Invest. 2008 Mar;38(3):197-200. doi: 10.1111/j.1365-2362.2008.01907.x. PMID 18257783
- [Background] Weschta M, Deutschle T, Riechelmann H. Nasal fractional exhaled nitric oxide analysis with a novel hand-held device. Rhinology. 2008 Mar;46(1):23-7. PMID 18444488
- [Background] Marthin JK, Nielsen KG. Hand-held tidal breathing nasal nitric oxide measurement--a promising targeted case-finding tool for the diagnosis of primary ciliary dyskinesia. PLoS One. 2013;8(2):e57262. doi: 10.1371/journal.pone.0057262. Epub 2013 Feb 20. PMID 23437356
- [Background] Montella S, Alving K, Maniscalco M, Sofia M, De Stefano S, Raia V, Santamaria F. Measurement of nasal nitric oxide by hand-held and stationary devices. Eur J Clin Invest. 2011 Oct;41(10):1063-70. doi: 10.1111/j.1365-2362.2011.02501.x. Epub 2011 Mar 17. PMID 21413977